CLINICAL TRIAL: NCT01686269
Title: Mobilization of Endothelial Progenitor Cells in Patients With Coronary Artery Bypass Surgery
Brief Title: Endothelial Progenitor Cells
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FEMH-95-C-018
Record Dates: First submitted 2009-02-06; First posted 2012-09-18 (Estimated); Last update posted 2012-09-18 (Estimated); Status verified 2007-01

CONDITIONS: Coronary Artery Disease
Keywords: Endothelial progenitor cell; coronary artery bypass
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: blood collecting

SUMMARY:
Vascular stenosis as a result of neointimal hyperplasia is a major clinical problem that has an impact on multiple and diverse disciplines, including cardiology (coronary restenosis), cardiothoracic and vascular surgery (saphenous vein and polytetrafluoroethylene [PTFE] graft failure), neurology (carotid stenosis), nephrology (dialysis access dysfunction), and transplant medicine (chronic allograft rejection in hearts and kidneys). [1] In marked contrast to the deleterious effects of smooth muscle progenitor cells on neointimal hyperplasia, circulating endothelial progenitor cells (EPCs) are believed to play an important role in vascular repair and in the inhibition of neointimal hyperplasia. [2] Endothelial progenitor cells (EPCs) circulate in adult peripheral blood and contribute to neovascularization. Satoshi et al. have demonstrated that lineage-committed EPCs and CD34-positive mononuclear cells, their putative precursors, are mobilized during an acute ischemic event in humans. [3] Reduced levels of circulating EPCs independently predict atherosclerotic disease progression, thus supporting an important role for endogenous vascular repair to modulate the clinical course of coronary artery disease. [4] These observations prompt the hypothesis that circulating EPCs may provide an endogenous repair mechanism to counteract surgery-induced endothelial cell injury and to replace dysfunctional endothelium perioperatively. Therefore, the investigators examined whether levels of circulating EPCs correlate with time course and outcomes of coronary artery bypass surgery to establish a clinical role of endogenous endothelial repair mediated by circulating EPCs.

ELIGIBILITY:
Inclusion Criteria:

* age from 18 to 85 years
* signed written informed consent
* angiographically documented coronary artery disease and indicated for coronary artery bypass surgery

Exclusion Criteria:

* clinical or biochemical evidence for the presence of concomitant inflammatory disease
* chronic renal insufficiency (serum creatinine > 1.4 mmol/L)
* impaired left ventricular ejection fraction (< 45%)
* autoimmune or malignant disease
* thrombocytopenia (< 100 000/L)
* anemia (hemoglobin < 8.5 g/dL)
* inability to understand the consent form
* previous coronary bypass surgery
* severe peripheral arterial occlusive disease or atrial fibrillation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2007-03

CONTACTS AND LOCATIONS:
Overall Officials: Kuan-Ming Chiu, MD, Study Director — Far Eastern Memorial Hospital
Locations (1):
- Far Eastern Memorial Hospital, Taipei, Taiwan